CLINICAL TRIAL: NCT00049023
Title: A Phase I, Open Label, Maximum Tolerated Dose-Finding Study to Evaluate the Safety and Tolerability of 90Y-DOTA-tyr3-Octreotide Administered by Intravenous Infusion to Children With Refractory Somatostatin-Receptor Positive Tumors
Brief Title: Radiolabeled Octreotide in Treating Children With Advanced or Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: O'Dorisio, M S (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, O'Dorisio, M S, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200008086; UIHC-200008086; NCI-V02-1710
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Brain and Central Nervous System Tumors; Gastrointestinal Carcinoid Tumor; Islet Cell Tumor; Neuroblastoma; Pheochromocytoma; Sarcoma; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: childhood grade III meningioma; disseminated neuroblastoma; localized unresectable neuroblastoma; metastatic pheochromocytoma; metastatic Ewing sarcoma/peripheral primitive neuroectodermal tumor; recurrent childhood brain tumor; recurrent childhood medulloblastoma; recurrent neuroblastoma; recurrent pheochromocytoma; recurrent Ewing sarcoma/peripheral primitive neuroectodermal tumor; regional neuroblastoma; regional pheochromocytoma; unspecified childhood solid tumor, protocol specific; recurrent childhood ependymoma; childhood infratentorial ependymoma; childhood supratentorial ependymoma; recurrent islet cell carcinoma; gastrinoma; insulinoma; metastatic gastrointestinal carcinoid tumor; recurrent gastrointestinal carcinoid tumor; regional gastrointestinal carcinoid tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Adenoma, Islet Cell; Neuroblastoma; Pheochromocytoma; Sarcoma; Neuroectodermal Tumors, Primitive, Peripheral; Medulloblastoma; Familial ependymoma; Carcinoma, Islet Cell; Gastrinoma; Insulinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 90Y-DOTA-tyr3-OCTREOTIDE (Experimental): Dose escalation will proceed so that the single-cycle and three-cycle maximum tolerated doses of 90Y-DOTA-tyr3-Octreotide can be determined. The initial dose of 90Y-DOTA-tyr3-Octreotide to be administered is 30 mCi/m2 in each of three cycles. Dose escalation will proceed in 10 mCi/m2 intervals and will be permitted for the next cohort of subjects pending completion of Cycle 3 by 2 members of the previous cohort with no DLTs. A DLT is defined as a Grade 3 renal toxicity, Grade 4 bone marrow toxicity, or any other Grade 3 toxicity whether or not related to study drug and regardless of duration. Lymphopenia will not be used to define a DLT.
  Interventions: Radiation: 90Y-DOTA-tyr3-OCTREOTIDE

INTERVENTIONS:
Radiation: 90Y-DOTA-tyr3-OCTREOTIDE

SUMMARY:
RATIONALE: Radiolabeled octreotide can locate tumor cells and deliver radioactive tumor-killing substances to them without harming normal cells.

PURPOSE: This phase I trial is to study the safety and effectiveness of radiolabeled octreotide in treating children who have advanced or refractory solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of yttrium Y 90-DOTA-tyr3-octreotide in children with advanced or refractory somatostatin receptor-positive tumors.
* Determine the short-term and long-term safety and the serious adverse-event profiles of this drug in these patients.
* Determine any potential antitumor effect of this drug in these patients.
* Correlate level of somatostatin receptor type 2 expression with response in patients treated with this drug.

OUTLINE: This is a dose-escalation study.

Patients receive yttrium Y 90-DOTA-tyr3-octreotide IV over 5-10 minutes on day 1. Treatment repeats every 6 weeks for up to 3 courses in the absence of unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of yttrium Y 90-DOTA-tyr3-octreotide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 6 patients experience dose-limiting toxicity.

Patients are followed weekly after each treatment course, 6 weeks after the last course, and then every 6 months thereafter for life.

PROJECTED ACCRUAL: Approximately 25-35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed malignant neoplasm

  * Not amenable to standard therapy or has failed existing first- and second-line therapies
* Tumor positive for somatostatin receptors by OctreoScan within the past 4 weeks
* At least 1 measurable lesion

  * Lesions that have been previously irradiated must demonstrate progression since radiation
  * At least 1 measurable somatostatin receptor-positive lesion that has not been irradiated within the past 4 weeks AND has not had full craniospinal radiation within the past 3 months
* Bone marrow with at least 40% cellularity OR at least 20% cellularity with one million CD34+ stem cells/kg stored
* No diffuse bone marrow involvement by OctreoScan scintigraphy

PATIENT CHARACTERISTICS:

Age

* 2 to 25

Performance status

* COG 0-2 OR
* Karnofsky 60-100% OR
* Lansky 60-100%

Life expectancy

* 2-12 months

Hematopoietic

* See Disease Characteristics
* Absolute neutrophil count at least 1,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin less than 1.5 times normal
* AST and ALT less than 2.5 times upper limit of normal

Renal

* Creatinine no greater than 1 mg/dL (children less than 5 years of age)
* Creatinine less than 1.2 mg/dL (children 5 to 10 years of age)
* Creatinine less than 1.7 mg/dL (children over 10 years of age) AND
* Glomerular filtration rate at least 80 mL/min/m^2

Cardiovascular

* Shortening fraction at least 28% by echocardiogram
* Ejection fraction at least 50% by bi-plane method of echocardiogram
* No prior congestive heart failure unless ejection fraction at least 40%
* No unstable angina pectoris
* No cardiac arrhythmia
* No symptomatic congestive heart failure

Other

* No other concurrent malignancy
* No other significant uncontrolled medical, psychiatric, or surgical condition that would preclude study compliance
* No antibodies to yttrium Y 90-DOTA-tyr3-octreotide or octreotide
* No prior allergic reactions to compounds of similar chemical or biologic composition to yttrium Y 90-DOTA-tyr3-octreotide
* No ongoing or active infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)

Endocrine therapy

* More than 28 days since prior long-acting somatostatin analogues
* No concurrent somatostatin analogues 12 hours before or 12 hours after study drug administration
* Concurrent hormonal therapy (other than somatostatin analogue) allowed provided patient received hormonal therapy for at least 2 months and has stable disease or progressive disease

Radiotherapy

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy
* No prior radiotherapy to 25% or more of bone marrow
* No prior external beam radiotherapy to both kidneys (scatter doses of less than 500 cGy to a single kidney or radiation to less than 50% of a single kidney is allowed)

Surgery

* At least 4 weeks since prior surgery

Other

* Recovered from prior therapy
* At least 4 weeks since prior investigational drugs
* No other concurrent approved or investigational anti-neoplastic therapies except for bisphosphonates
* No concurrent combination antiretroviral therapy for HIV-positive patients

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2002-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Establish the three-cycle maximum-tolerated dose of 90Y-DOTA-tyr3-Octreotide | 6 weeks per cycle
  Establish the three-cycle maximum-tolerated dose of 90Y-DOTA-tyr3-Octreotide administered by intravenous infusion to children with refractory somatostatin-receptor positive tumors based upon the 6 week/cycle dose-limiting-toxicity profile.
Evaluate the short term and long term safety (mild/moderate/severe/life-threatening adverse events, premature discontinuations and serious adverse events) | short term (6 weeks/cycle); long term (4-6 mos./cycle)
  2. Evaluate the short-term (6 weeks/cycle) and long term (4-6 months) safety (mild/moderate/severe/life-threatening adverse events, premature discontinuations and serious adverse events) serious adverse event profile of three-cycles of 90Y-DOTA-tyr3-Octreotide administered by intravenous infusion to children with refractory somatostatin-receptor positive tumors.

CONTACTS AND LOCATIONS:
Overall Officials: M. Sue O'Dorisio, MD, PhD, Study Chair — Holden Comprehensive Cancer Center
Locations (1):
- Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa, United States

REFERENCES:
- [Result] Menda Y, O'Dorisio MS, Kao S, Khanna G, Michael S, Connolly M, Babich J, O'Dorisio T, Bushnell D, Madsen M. Phase I trial of 90Y-DOTATOC therapy in children and young adults with refractory solid tumors that express somatostatin receptors. J Nucl Med. 2010 Oct;51(10):1524-31. doi: 10.2967/jnumed.110.075226. Epub 2010 Sep 16. PMID 20847174